CLINICAL TRIAL: NCT01238874
Title: Latin America Cardiac Resynchronization Therapy Study
Acronym: LatAmCRT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medtronic Latin America (Industry)
Responsible Party: Hugo Fagioli/Clinical Research Director, Medtronic Latin America
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LA CRT Study
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Heart Failure.
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

ARMS (1):
- No intervention (No Intervention): Mostly observational study with 1 patient global assessment.
  Interventions: Device: Cardiac Resynchronization Therapy

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy — All market-approved Medtronic CRT-D and CRT-P devices will be used in this study. All eligible devices are commercially released and will be used within their intended use per device labeling. The study may include future market-approved devices as they become commercially available. All market-approved leads may be used in the study. Epicardial leads may be used in the study.

SUMMARY:
The Latin America CRT Study is a prospective, multicenter, interventional post-market release study conducted in Latin America. The geography includes Puerto Rico and the Caribbean, Mexico and Central America, and South America.

DETAILED DESCRIPTION:
The purpose of this study is to provide local evidence regarding Cardiac Resynchronization Therapy (CRT), in both pacing and defibrillation devices across Latin America. The primary objective will focus on changes in left ventricular heart size and function measurements in subjects receiving CRT therapy. The following additional parameters will also be collected:

* Data on referral patterns in Latin America;
* Data on device implant (including delivery system, device information, and lead information);
* Clinical data on subject outcomes and changes (improved, unchanged, or worsened) in heart failure status as assessed by heart failure (HF) hospitalizations, New York Heart Association (NYHA) class, mortality, and Quality of Life (QOL) measured by the Patient Global Assessment;

ELIGIBILITY:
Inclusion Criteria: Implant of new CRT-D or CRT-P device (first-time implant), ACC/AHA/HRS/ESC guidelines for implant, NYHA Class II, III or IV, QRS duration >120 ms, LVEF < 35%, Receiving optimal medical/drug therapy, Able to give written informed consent, Are > 21 years of age, Must be able to return for follow-up visits as required, Are not pregnant or do not plan to get pregnant within the next 6 months, Have no physical limitations to perform Echo studies

Exclusion Criteria: Previous or existing CRT system implanted, Unwilling or unable to comply with specified follow-up schedule, Enrolled or intending to participate in another device study during the course of this study that requires specific treatment or device programming, Medical condition that may limit life expectancy to < 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Measure heart size and function changes as assessed by Doppler echocardiogram (Echo). | 6 Months
  Measure heart size and function changes as assessed by Doppler echocardiogram (Echo).

SECONDARY OUTCOMES:
referral patterns; Report on device implant; Analyze subject clinical status as it pertains to heart failure (HF) hospitalizations, changes in NYHA class, mortality and QOL (Patient Global Assessment); | 6 Months
  referral patterns; Report on device implant; Analyze subject clinical status as it pertains to heart failure (HF) hospitalizations, changes in NYHA class, mortality and QOL (Patient Global Assessment);

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - Hospital Angeles Tijuana, Tijuana, Estado de Baja California
  - Hospital Angeles Leon, León, Guanajuato